CLINICAL TRIAL: NCT01073384
Title: A Phase 1/2 Study to Evaluate Escalating Doses of SGX201 [Delayed Release Oral Beclomethasone Dipropionate (BDP)] for Prevention of Signs and Symptoms of Acute Enteritis in Patients With Rectal Cancer Treated With Combined Chemotherapy and Radiation Therapy
Brief Title: A Dose Ranging Study of Delayed Release Beclomethasone for Prevention of Acute Enteritis in Patients With Rectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Soligenix (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BDP-ENT-01; 1R43CA141968-01 (NIH)
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Enteritis
MeSH Terms: conditions — Enteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- BDP 3 mg (Experimental): 1 mg TID
  Interventions: Drug: SGX201 (delayed release beclomethasone 17,21-dipropionate)
- BDP 6 mg (Experimental): 2 mg TID
  Interventions: Drug: SGX201 (delayed release beclomethasone 17,21-dipropionate)
- BDP 9 mg (Experimental): 3 mg TID
  Interventions: Drug: SGX201 (delayed release beclomethasone 17,21-dipropionate)
- BDP 12 mg (Experimental): 4 mg TID
  Interventions: Drug: SGX201 (delayed release beclomethasone 17,21-dipropionate)

INTERVENTIONS:
Drug: SGX201 (delayed release beclomethasone 17,21-dipropionate) — Delayed release beclomethasone 17,21-dipropionate before the first administration of radiation therapy continuing for 7 days after the end of radiation therapy.
  Other Names: beclomethasone 17,21-dipropionate; 17,-21 BDP

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of four doses of SGX201 in subjects with rectal cancer treated with concurrent radiation and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary rectal cancer
* Planned course of conventional neoadjuvant radiation therapy before surgery
* Scheduled to receive chemotherapy
* >/= 18 years of age
* Negative pregnancy test

Exclusion Criteria:

* History of acute or chronic regional enteritis or inflammatory bowel disease
* Stool incontinence
* Uncontrollable diarrhea
* Abdominal-perineal resection or other surgery leaving patient without a functioning rectum
* Patients using colostomy or ileostomy
* Liver function tests > 3x upper limit of normal, or bilirubin test result > 1.5 the upper limit of normal
* Calculated creatinine clearance <60 mL/minute
* Planned hyperfractionated or split course radiation
* Planned brachytherapy prior to completion of all external beam radiation therapy
* Prior pelvic RT
* An on-going infection
* ECOG score >/= 3
* Leukopenia <2,000 WBC/mm3 or Hg <10.5 g/dL
* Participation in an investigational drug trial within the previous 30 days
* Patients with a medical condition that would interfere with study compliance
* Known hypersensitivity to 5-FU or capecitabine
* Anticipated inability to tolerate oral administration of SGX201
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Preliminary Efficacy | One day prior to and 7 days after radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Horgan, MD, Principal Investigator — Soligenix
Locations (2):
- United States (2):
  - Northwestern University Medical Center, Chicago, Illinois
  - Boston University, Boston, Massachusetts

REFERENCES:
- See also: Sponsor — http://www.soligenix.com